CLINICAL TRIAL: NCT06281080
Title: First-in-Human Trial of a Novel Endoluminal Robotic System for En-Bloc Resection of Bladder Tumours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Agilis Robotics Limited (Unknown)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE2023.589-T
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Patients underwent En-Bloc Resection of Bladder Tumours using Agilis Robotic System.
  Interventions: Procedure: En-Bloc Resection of Bladder Tumours

INTERVENTIONS:
Procedure: En-Bloc Resection of Bladder Tumours — Patients underwent En-Bloc Resection of Bladder Tumours using Agilis Robotic System.

SUMMARY:
This is a prospective, single-arm study to evaluate the feasibility and safety of performing transurethral en-bloc resection of bladder tumours using the Zenith robotic system.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years
2. Body mass index <35 kg/m2
3. Bladder tumour located <3 cm in size; clinically non-muscle invasive bladder tumour
4. Clinically indicated for en-bloc resection.
5. Willingness to participate as demonstrated by giving informed consent

Exclusion Criteria:

1. Presence of endoscopic or imaging signs of detrusor muscle invasion
2. Contraindication to general anaesthesia / spinal anaesthesia
3. ASA > 2 patients
4. Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic intervention
5. Untreated active infection
6. Un-corrected coagulopathy
7. Presence of another malignancy or distant metastasis
8. Emergency surgery
9. Vulnerable population (e.g. mentally disabled, pregnant)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Successful en-bloc tumour resection by the robotic system | During the operation
  The number of cases completed the intervention by robotic system

SECONDARY OUTCOMES:
Dissection time and speed | During operation
  Time required for submucosal dissection from the first cut
Total procedure time | During operation
  Time from insertion of the robotic system into urethra until removal of the specimen from the body
Surgeon Console time | During operation
  From the time start of any procedure to completion of urethral catheter insertion
Presence of detrusor muscle in specimen | During operation
  Presence of detrusor muscle in specimen
Resection Margin | During operation
  Number of subject with Negative resection margin
Intra-operative bladder perforation event | During operation
  Number of subject
Post-operative complications | Within 90 days after the study intervention
  Complication is defined according to the Clavien-Dindo Classification
Need of bladder irrigation | Within 30 days after the study intervention.
  Number of subject
Residual tumour or upstaging of tumour after second look TURBT | Within 30 days after the study intervention.
  Number of subject

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maurice MJ, Vricella GJ, MacLennan G, Buehner P, Ponsky LE. Endoscopic snare resection of bladder tumors: evaluation of an alternative technique for bladder tumor resection. J Endourol. 2012 Jun;26(6):614-7. doi: 10.1089/end.2011.0587. Epub 2012 May 3. PMID 22390750
- [Background] Gontero P, Sylvester R, Pisano F, Joniau S, Vander Eeckt K, Serretta V, Larre S, Di Stasi S, Van Rhijn B, Witjes AJ, Grotenhuis AJ, Kiemeney LA, Colombo R, Briganti A, Babjuk M, Malmstrom PU, Oderda M, Irani J, Malats N, Baniel J, Mano R, Cai T, Cha EK, Ardelt P, Varkarakis J, Bartoletti R, Spahn M, Johansson R, Frea B, Soukup V, Xylinas E, Dalbagni G, Karnes RJ, Shariat SF, Palou J. Prognostic factors and risk groups in T1G3 non-muscle-invasive bladder cancer patients initially treated with Bacillus Calmette-Guerin: results of a retrospective multicenter study of 2451 patients. Eur Urol. 2015 Jan;67(1):74-82. doi: 10.1016/j.eururo.2014.06.040. Epub 2014 Jul 16. PMID 25043942
- [Background] Ukai R, Kawashita E, Ikeda H. A new technique for transurethral resection of superficial bladder tumor in 1 piece. J Urol. 2000 Mar;163(3):878-9. PMID 10687997
- [Background] Paciotti M, Casale P, Colombo P, Fasulo V, Saita A, Lughezzani G, Contieri R, Buffi NM, Lazzeri M, Guazzoni G, Hurle R. Long-term Follow-up After En Bloc Transurethral Resection of Non-muscle-invasive Bladder Cancer: Results from a Single-center Experience. Eur Urol Open Sci. 2021 Feb 24;26:64-71. doi: 10.1016/j.euros.2021.01.015. eCollection 2021 Apr. PMID 34337509
- [Background] Cheng YY, Sun Y, Li J, Liang L, Zou TJ, Qu WX, Jiang YZ, Ren W, Du C, Du SK, Zhao WC. Transurethral endoscopic submucosal en bloc dissection for nonmuscle invasive bladder cancer: A comparison study of HybridKnife-assisted versus conventional dissection technique. J Cancer Res Ther. 2018;14(7):1606-1612. doi: 10.4103/jcrt.JCRT_786_17. PMID 30589047
- [Background] Zhang KY, Xing JC, Li W, Wu Z, Chen B, Bai DY. A novel transurethral resection technique for superficial bladder tumor: retrograde en bloc resection. World J Surg Oncol. 2017 Jul 6;15(1):125. doi: 10.1186/s12957-017-1192-6. PMID 28683751
- [Background] Teoh JY, MacLennan S, Chan VW, Miki J, Lee HY, Chiong E, Lee LS, Wei Y, Yuan Y, Yu CP, Chow WK, Poon DM, Chan R, Lai F, Ng CF, Breda A, Kramer MW, Malavaud B, Mostafid H, Herrmann T, Babjuk M. An International Collaborative Consensus Statement on En Bloc Resection of Bladder Tumour Incorporating Two Systematic Reviews, a Two-round Delphi Survey, and a Consensus Meeting. Eur Urol. 2020 Oct;78(4):546-569. doi: 10.1016/j.eururo.2020.04.059. Epub 2020 May 8. PMID 32389447
- [Background] Hurle R, Lazzeri M, Colombo P, Buffi N, Morenghi E, Peschechera R, Castaldo L, Pasini L, Casale P, Seveso M, Zandegiacomo S, Taverna G, Benetti A, Lughezzani G, Fiorini G, Guazzoni G. "En Bloc" Resection of Nonmuscle Invasive Bladder Cancer: A Prospective Single-center Study. Urology. 2016 Apr;90:126-30. doi: 10.1016/j.urology.2016.01.004. Epub 2016 Jan 14. PMID 26776561
- [Background] Teoh JY, Mayor N, Li KM, Lo KL, Ng CF, Mostafid H. En-bloc resection of bladder tumour as primary treatment for patients with non-muscle-invasive bladder cancer: routine implementation in a multi-centre setting. World J Urol. 2021 Sep;39(9):3353-3358. doi: 10.1007/s00345-021-03675-9. Epub 2021 Mar 28. PMID 33774705
- [Background] McCulloch P, Altman DG, Campbell WB, Flum DR, Glasziou P, Marshall JC, Nicholl J; Balliol Collaboration; Aronson JK, Barkun JS, Blazeby JM, Boutron IC, Campbell WB, Clavien PA, Cook JA, Ergina PL, Feldman LS, Flum DR, Maddern GJ, Nicholl J, Reeves BC, Seiler CM, Strasberg SM, Meakins JL, Ashby D, Black N, Bunker J, Burton M, Campbell M, Chalkidou K, Chalmers I, de Leval M, Deeks J, Ergina PL, Grant A, Gray M, Greenhalgh R, Jenicek M, Kehoe S, Lilford R, Littlejohns P, Loke Y, Madhock R, McPherson K, Meakins J, Rothwell P, Summerskill B, Taggart D, Tekkis P, Thompson M, Treasure T, Trohler U, Vandenbroucke J. No surgical innovation without evaluation: the IDEAL recommendations. Lancet. 2009 Sep 26;374(9695):1105-12. doi: 10.1016/S0140-6736(09)61116-8. PMID 19782876
- [Background] McCulloch P, Cook JA, Altman DG, Heneghan C, Diener MK; IDEAL Group. IDEAL framework for surgical innovation 1: the idea and development stages. BMJ. 2013 Jun 18;346:f3012. doi: 10.1136/bmj.f3012. PMID 23778427
- [Background] Bilbro NA, Hirst A, Paez A, Vasey B, Pufulete M, Sedrakyan A, McCulloch P; IDEAL Collaboration Reporting Guidelines Working Group. The IDEAL Reporting Guidelines: A Delphi Consensus Statement Stage Specific Recommendations for Reporting the Evaluation of Surgical Innovation. Ann Surg. 2021 Jan 1;273(1):82-85. doi: 10.1097/SLA.0000000000004180. PMID 32649459